CLINICAL TRIAL: NCT00085826
Title: A Phase III, Randomized, Double-Blind, Multi-Center Study of the Efficacy of Taxotere (Docetaxel) in Combination With Aptosyn (Exisulind) Versus Taxotere (Docetaxel) and Placebo in Non-Small Cell Lung Cancer (NSCLC) Patients After Failure of Prior Platinum-Based Chemotherapy
Brief Title: A Phase III Study of the Efficacy of Taxotere/Aptosyn Versus Taxotere/Placebo in Non-Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 028; NCT00021411 (obsolete NCT alias); NCT00036322 (obsolete NCT alias)
Record Dates: First submitted 2004-06-15; First posted 2004-06-17 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer; NSCLC; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — sulindac sulfone

INTERVENTIONS:
Drug: Exisulind

SUMMARY:
Taxotere has been approved by the FDA and is considered a standard treatment for patients with lung cancer who have failed prior platinum-containing regimens. The main purpose of this research study is to determine if Aptosyn, when given in combination with Taxotere, will result in prolonged survival when compared to Taxotere alone.

This study will also help determine tumor response rates, and the safety profile of Aptosyn in combination with Taxotere.

This study has been completed and a publication is pending.

ELIGIBILITY:
Exclusion Criteria:

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2001-04; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (110):
  - Birmingham Hematology Oncology Associates, Birmingham, Alabama
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Northern Arizona Hematology and Oncology Associates, Flagstaff, Arizona
  - Hematology & Oncology Associates, Phoenix, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Arkansas Oncology Associates, PA, Little Rock, Arkansas
  - Pacific Coast Hematology/Oncology Medical Group, Inc., Fountain Valley, California
  - California Cancer Care, Inc., Greenbrae, California
  - Scripps Cancer Center, San Diego, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Rocky Mountain Cancer Center, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - RMCC, Denver, Colorado
  - 12. Rocky Mountain Cancer Centers-Englewood, Englewood, Colorado
  - Rocky Mountain Cancer Centers, Englewood, Colorado
  - Rocky Mountain Cancer Centers, Fort Collins, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Comprehensive Cancer Care Specialists at Boca Raton, Boca Raton, Florida
  - North Florida Hematology & Oncology Association, Jacksonville, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - South Florida Oncology & Hematology Consultants, Lauderhill, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Cancer Centers of Florida, Orlando, Florida
  - Lauderhill Lakes, Plantation, Florida
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Northwest Medical Specialists, PC, Niles, Illinois
  - Onc/Hem Associates of Central Illinois, Peoria, Illinois
  - Hematology Oncology Associates of Illinois, Skokie, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Iowa Cancer Care, PLC, Cedar Rapids, Iowa
  - Iowa Oncology Associates, Cedar Rapids, Iowa
  - Central Maryland Oncology Center, Columbia, Maryland
  - Central Maryland Oncology Group, Towson, Maryland
  - Impath Predictive Oncology, Franklin, Massachusetts
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Minnesota Oncology Hematology, PA, Saint Paul, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri
  - The Center for Cancer Care & Research, St Louis, Missouri
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - New Mexico Cancer Center Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, PC, Albany, New York
  - New York Oncology Hematology, Albany, New York
  - HemOnCare, PC, Brooklyn, New York
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Cancer Research of Long Island, Great Neck, New York
  - Interlakes Oncology & Hematology, P.C., Rochester, New York
  - Asheville Hematology & Oncology Associates, PA, Asheville, North Carolina
  - Raleigh Hematology Oncology Clini, Cary, North Carolina
  - Regional Hamatology Oncology Associates, Durham, North Carolina
  - Northeastern Carolina Hematology & Oncology, PA, Hickory, North Carolina
  - Raleigh Hematology Oncology Clinic, Raleigh, North Carolina
  - Piedmont Hematology Onccology Associates, P.A., Winston-Salem, North Carolina
  - Dayton Oncology/Hematology, PA, Kettering, Ohio
  - Cancer Care Associates - Baptist Campus, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Hematology & Oncolgy Assoc of NE PA, Dunmore, Pennsylvania
  - Medical Oncology Associates of Wymoning Valley, PC, Kingston, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple Cancer Center, Philadelphia, Pennsylvania
  - Oncology-Hematology Associates, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Texas Oncology, PA, Abilene, Texas
  - Texas Oncology, P.A, Arlington, Texas
  - South Austin Cancer Center, Austin, Texas
  - Mamie McFadden Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - US Oncology Research, Dallas, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Onclology, PA, Dallas, Texas
  - The Texas Cancer Center - Dallas Southwest, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Texoma Cancer Center, Denison, Texas
  - Texas Cancer Center, Fort Worth, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - San Antonio Tumor and Blood Clinic, Fredicksburg, Texas
  - Texas Oncology, PA, Garland, Texas
  - Texas Oncology, PA, Houston, Texas
  - Texas Oncology, PA, Irving, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - an Antonio Tumor and Blood Clinic, San Antonio, Texas
  - Hematology Oncology Associates of South Texas, San Antonio, Texas
  - San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer Care & Research Center, Waco, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Fairfax Northern Virginia Hematology-Oncology, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates of South West Virginia, Inc., Salem, Virginia
  - Puget Sound Cancer Centers, Edmonds, Washington
  - Ranier Oncology Professional Services, Puyallup, Washington
  - Washington Cancer Center, P.C.Puget Sound Cancer Cente, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - MultiCare Health System, Tacoma, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin